CLINICAL TRIAL: NCT03448367
Title: FreeStyle Libre Flash Glucose Monitoring System Post Approval Study for Pediatric Patients
Status: Terminated | Type: Observational
Why Stopped: Due to lower than anticipated enrollment
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-PMS-17168-002
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- SMBG/FreeStyle Libre: During the intervention phase, subjects will use FreeStyle Libre Flash Glucose Monitoring System for 6 months to managed their diabetes.
  Interventions: Device: FreeStyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will utilize capillary SMBG for managing diabetes for 6 months (control phase) followed by diabetes management using FreeStyle Libre for 6 months (intervention phase).

SUMMARY:
This is a prospective, multi-center, non-randomized, single-arm, post-approval study of the FreeStyle Libre Flash Glucose Monitoring System intended to characterize the safety of the Libre Flash Glucose Monitoring System when used in pediatric patients with diabetes.

DETAILED DESCRIPTION:
Up to 400 pediatric subjects aged 4-17 years with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes, will be enrolled to obtain at least 314 subjects who complete the final visit. Subjects and/or their caregivers will utilize capillary SMBG for managing diabetes for 6 months (control phase) followed by diabetes management using FreeStyle Libre for 6 months (intervention phase). Subjects and/or their caregivers will maintain a diary/log book of Adverse Events during each phase. Assessment of Adverse Events will occur via self reporting at each monthly visit and/or phone call.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 4 - 17 years of age.
* Subject must have a diagnosis of type 1 or type 2 diabetes mellitus for at least 3 months prior to enrollment.
* Subject is currently using SMBG for managing their diabetes.
* Subject and/or caregiver must be able to read and understand English .
* In the investigator's opinion, the subject and/or caregiver must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Subject and/or caregiver must have access to an internet connected computer for uploading data from the blood glucose meter and FreeStyle Libre system.
* Subject must have an overnight companion (caregiver 18 years or older) present in the same home during participation of the study.
* Subject and/or parent or guardian must be willing and able to provide written signed and dated informed consent and assent when appropriate.

Exclusion Criteria:

* Subject and/or caregiver is a member of the Site Staff.
* Subject is currently using or has previously used a continuous glucose monitoring system for managing their diabetes
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is known to be pregnant or is attempting to become pregnant at the time of enrollment.
* Subject is on dialysis at the time of enrollment.
* Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff.
* Subject currently is participating in another clinical trial.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric subjects aged 4-17 years and older with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes. At least 50% of the study population will be age 4-12 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Safety of the FreeStyle Libre Flash Glucose Monitoring System | Approximately one year per subject.
  The study is designed to characterize the safety of the FreeStyle Libre Flash Glucose Monitoring System when used in the pediatric patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (4):
- United States (4):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No